CLINICAL TRIAL: NCT00283751
Title: Comparison of Efficacy and Safety of Insulin Detemir and Insulin Glargine as Add-on to Current Oral Antidiabetic Drugs in Subjects With Type 2 Diabetes
Brief Title: Comparison of Insulin Detemir or Insulin Glargine as Add on to Oral Antidiabetic Drugs in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1373
Record Dates: First submitted 2006-01-27; First posted 2006-01-30 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin detemir
Drug: insulin glargine

SUMMARY:
This trial is conducted in Europe and the United States of America (USA). The aim of the trial is to test if Insulin Detemir as add-on to current Oral Antidiabetic Drug treatment is at least as effective as Insulin Glargine as add-on to current Oral Antidiabetic Drug treatment in reducing HbA1c in patients with Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes for more than 12 months, and no previous insulin treatment
* Oral Antidiabetic Drug treatment for at least 4 months
* Body Mass Index (BMI) less than 40 kg/m2
* HbA1c 7.5-10.0%

Exclusion Criteria:

* Current or previous treatment with thiazolidinediones within the last 6 months
* Oral Antidiabetic Drug treatment with combination of three or more Oral Antidiabetic Drugs within the last 6 months
* Proliferative retinopathy or maculopathy
* Known hypoglycaemia unawareness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 583 (Actual)
Dates: Start 2003-03; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 52 weeks

SECONDARY OUTCOMES:
Insulin antibodies
Incident of hypoglycaemic episodes and adverse events
Plasma glucose profiles
Change in body weight

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (88):
- United States (19):
  - Novo Nordisk Investigational Site, Greenbrae, California
  - Novo Nordisk Investigational Site, La Mesa, California
  - Novo Nordisk Investigational Site, West Palm Beach, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Springfield, Illinois
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Chesterfield, Missouri
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Lincoln, Nebraska
  - Novo Nordisk Investigational Site, Pleasantville, New Jersey
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Kettering, Ohio
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Mt. Pleasant, South Carolina
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Warrenton, Virginia
  - Novo Nordisk Investigational Site, Seattle, Washington
- Austria (6):
  - Novo Nordisk Investigational Site, Ebreichsdorf
  - Novo Nordisk Investigational Site, Gratwein
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Neunkirchen
  - Novo Nordisk Investigational Site, Vienna
  - Novo Nordisk Investigational Site, Wolfsberg
- Belgium (5):
  - Novo Nordisk Investigational Site, Bonheiden
  - Novo Nordisk Investigational Site, Brussels
  - Novo Nordisk Investigational Site, Edegem
  - Novo Nordisk Investigational Site, Ghent
  - Novo Nordisk Investigational Site, Leuven
- France (12):
  - Novo Nordisk Investigational Site, Besançon
  - Novo Nordisk Investigational Site, Bondy
  - Novo Nordisk Investigational Site, Grenoble
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Lyon
  - Novo Nordisk Investigational Site, Nantes
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Nîmes
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Poitiers
  - Novo Nordisk Investigational Site, Strasbourg
  - Novo Nordisk Investigational Site, Toulouse
- Germany (29):
  - Novo Nordisk Investigational Site, Bad Kreuznach
  - Novo Nordisk Investigational Site, Bad Mergentheim
  - Novo Nordisk Investigational Site, Bad Neuenahr-Ahrweiler
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Flensburg
  - Novo Nordisk Investigational Site, Frankfurt
  - Novo Nordisk Investigational Site, Freiburg im Breisgau
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Fürth
  - Novo Nordisk Investigational Site, Genthin
  - Novo Nordisk Investigational Site, Giessen
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Heidelberg
  - Novo Nordisk Investigational Site, Krefeld
  - Novo Nordisk Investigational Site, Ludwigshafen
  - Novo Nordisk Investigational Site, Marl
  - Novo Nordisk Investigational Site, München
  - Novo Nordisk Investigational Site, Neumünster
  - Novo Nordisk Investigational Site, Neuss
  - Novo Nordisk Investigational Site, Nuremberg
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Saarbrücken
  - Novo Nordisk Investigational Site, Saint Ingbert
  - Novo Nordisk Investigational Site, Schaafheim
  - Novo Nordisk Investigational Site, Schwabenheim
  - Novo Nordisk Investigational Site, Schwedt
  - Novo Nordisk Investigational Site, Völklingen
  - Novo Nordisk Investigational Site, Würzburg
- Novo Nordisk Investigational Site, Dublin, Ireland
- United Kingdom (16):
  - Novo Nordisk Investigational Site, Ayr
  - Novo Nordisk Investigational Site, Barnsley
  - Novo Nordisk Investigational Site, Bolton
  - Novo Nordisk Investigational Site, Bradford
  - Novo Nordisk Investigational Site, Church Village
  - Novo Nordisk Investigational Site, Cosham
  - Novo Nordisk Investigational Site, Dundee
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Harrow
  - Novo Nordisk Investigational Site, Leicester
  - Novo Nordisk Investigational Site, Livingstone
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Newcastle
  - Novo Nordisk Investigational Site, Poole
  - Novo Nordisk Investigational Site, Salford
  - Novo Nordisk Investigational Site, Swansea

REFERENCES:
- [Result] Rosenstock J, Davies M, Home PD, Larsen J, Koenen C, Schernthaner G. A randomised, 52-week, treat-to-target trial comparing insulin detemir with insulin glargine when administered as add-on to glucose-lowering drugs in insulin-naive people with type 2 diabetes. Diabetologia. 2008 Mar;51(3):408-16. doi: 10.1007/s00125-007-0911-x. Epub 2008 Jan 16. PMID 18204830
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com